CLINICAL TRIAL: NCT00773760
Title: Does mu Opioid Receptor (MOR) and Catechol-O-methyltransferase (COMT) Genes Polymorphism Correlate of Clinical Postoperative Pain and Response to Analgesics
Brief Title: MOR and COMT SNP Polymorphism and Pain
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: East Tallinn Central Hospital (Other)
Responsible Party: A.Veske PhD Director of Department of Gene Technology, TTU
Other Study IDs: ITK-1
Record Dates: First submitted 2008-10-15; First posted 2008-10-16 (Estimated); Last update posted 2009-08-06 (Estimated); Status verified 2009-08

CONDITIONS: Pain Relief
Keywords: opioids; COMT; SNP; analgesia; postoperative pain
MeSH Terms: conditions — Agnosia; Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- dosing
  Interventions: Other: SNP genotyping

INTERVENTIONS:
Other: SNP genotyping — Coded blood specimens will be transported to the Department of Gene Technology TTÜ and genotyping analysis will be performed. Lymphocytes will be isolated from blood specimens using Ficol-Paq gradients, and genomic DNA isolated using a salting-out procedure. Variants of the MOR gene and other genes of interests will be performed by DNA sequence analysis of PCR-amplified DNA, using primers located in flanking intron sequence. All methods proposed are currently in operation in the respective facilities.

SUMMARY:
Patients with certain polymorphism in the MOR and COMT genes will display differences in their response to analgesics.

DETAILED DESCRIPTION:
After tissue injury, there is great interindividual variability among patients in the amount of pain experienced (pain intensity and duration of pain) and in the degree of pain relief from analgesics. In experimental settings, Single Nucleotide Polymorphisms (SNP) at the MOR and COMT genes have been found to alter the response to opioids in in vitro models and in human.We will collect clinical data on one hundred patients undergoing surgery. We will obtain DNA extracted via PCR techniques from the patients' blood and we will identify SNPs at the mu opioid receptor and catechol-O-methyltransferase genes. We will analyze the data to search for correlation between clinical patterns of postoperative pain and opioid effects and SNPs.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* Give informed consent to participate in this study

Exclusion Criteria:

* Neurologic or psychiatric disease sufficient, in the clinical judgment of the investigator, to compromise informed consent or data collection
* ASA classification score 3 or above
* Patients with past or present history of substance abuse.
* Patients with a history of chronic pain requiring daily analgesic use for more then one month.
* Patients with a current diagnosis of anxiety or depression requiring medical treatment
* Patients allergic to morphine

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with prostate cancer
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2008-10; Primary Completion 2009-10 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Postoperative assessments include PCA use (e.g., number of patient demands, total morphine administered) in each 24-h interval during the 48-h study period - primary endpoint. | 48 hours

SECONDARY OUTCOMES:
No secondary outcome endpoint | no time frame

CONTACTS AND LOCATIONS:
Overall Officials: Yuri Kolesnikov, MD PhD, Study Director — ETCH
Locations (1):
- Yuri Kolesnikov MD PhD, Tallinn, Estonia

REFERENCES:
- See also: East Tallinn Central Hospital — http://www.itk.ee